CLINICAL TRIAL: NCT03833843
Title: Sudden Cardiac Death in Congenital Heart Diseases With a Systemic Right Ventricle
Brief Title: Sudden Cardiac Death in Systemic Right Ventricle
Acronym: STARSII
Status: Completed | Type: Observational
Sponsor: European Georges Pompidou Hospital (Other)
Collaborators: KU Leuven (Other); Erasmus Medical Center (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Centre Hospitalier Universitaire Vaudois (Other); University Hospital, Geneva (Other); Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Magalie Ladouceur, Principal Investigator, European Georges Pompidou Hospital
Other Study IDs: STARS
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Sudden Cardiac Death; Congenital Heart Disease; Transposition of Great Vessels
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Defects, Congenital; Transposition of Great Vessels | interventions — Diagnostic Imaging; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TGA
  Interventions: Diagnostic Test: imaging

INTERVENTIONS:
Diagnostic Test: imaging — ECG, Echocardiography and cardiac magnetic resonance imaging
  Other Names: Blood sample

SUMMARY:
In complete transposition of the great arteries (TGA) with previous atrial switch repair, and congenitally corrected transposition of the great arteries (ccTGA), the morphological right ventricle and its tricuspid valve continue to support the systemic circulation. This results in late complications including including sudden death.

This retrospective multicentric study aims to evaluate the prevalence of SCD in a contemporary population of patients with a systemic RV and identify specific risk factors for SCD and hemodynamically significant ventricular arrhythmia This registry records demographics, clinical, imaging data, electrophysiological and laboratory of patients with a sRV and a transposition of the great arteries Primary end points are defined by sudden cardiac death, near-miss sudden death, as well as sustained VT requiring defibrillation.

DETAILED DESCRIPTION:
1 Registry design

The registry is a retrospective multicentric registry that involves the collection of demographics, clinical, imaging data, electrophysiological and laboratory of patients with a sRV and a transposition of the great arteries (TGA or ccTGA).

Ethical or research committee approval should be obtained in each contributing center and all data will be collected retrospectively.

A minimum of 900 patients are expected to be registered.

Patient population Inclusion criteria: patients >16 years of age with a sRV and a transposition of the great arteries (TGA or ccTGA) with "two-ventricle circulation" under active follow-up between 2000 and 2018.

Exclusion criteria: CHD with univentricular heart physiology

2. Registry procedures

1. Design

   Data on all adult patients (>16 years of age) with sRV under active follow-up between January 1, 2000 and September 30, 2018 will be recorded. Baseline data, as well data of the last follow-up recorded during this period will be used.

   Parameters are chosen for inclusion in data collection on the basis of a review of sRV literature on single predictors of outcome The patients' medical records will be reviewed to collect demographic information, medical and surgical details

   The chosen parameters of patient past medical history to record include:
   * Type of TGA, TGA complexity, type of surgery, age at surgery, reoperation
   * Cardio-vascular events such as atrial arrhythmia, heart failure, pacemaker implantation
   * Performing electrophysiologic exploration and its results: normal or inducible sustained VT/VF, sinus node dysfunction, atrioventricular node dysfunction
   * 24H Holter ECG finding: sinus node disease, atrial arrhythmia, non-sustained VT, sustained VT
   * Notion of complete pregnancy (> 20 weeks of gestation)

   Baseline data will be taken at the first assessment as an adult (> 16 years old). They include variables from clinical status, 12-lead ECG, transthoracic echocardiography, CMR (if available), cardiopulmonary exercise test, and laboratory tests (if available). Detailed data are:
   * Clinical status: NYHA function class, syncope and palpitations.
   * Cardiac treatment
   * Electrocardiographic parameters, including rhythm assessment, heart rate, QRS duration, and QT interval manually collected
   * Echocardiographic parameters with visual sRVEF, tricuspid regurgitation grade, presence of pulmonary stenosis and baffle stenosis or leak. Only transthoracic echocardiography performed by experienced operators will be considered.
   * Measurements of oxygen consumption (VO2) during exercise test: peak oxygen consumption, VE/VCO2, peak blood pressure and peak heart rate.
   * If available, cardiac magnetic resonance imaging parameters, such as sRV volumes, sRV mass, sRVEF and presence of late gadolinium enhancement lesions.
   * If available, brain natriuretic peptide, with normal ranges provided by centers.

   Vital status at late follow-up during the study period (up to September 30, 2018) will be retrieved from national databases or patients' general practitioner records. Cardiac events such as heart failure, atrial arrhythmia, sustained ventricular tachycardia, death and cause of death will be reported.
2. Preservation and confidentiality of registry records Data collected at each investigational site will be entered in a local database. In this database, patient will be identifiable only by the investigator of the site. The data will be anonymized via the use of a unique number. This one will be created by a secure process called the function of occultation of the nominative information (FOIN). It will be impossible to find the identity of a patient from this number (irreversibility of encryption). The data will be anonymously transmitted to the main investigational site (Inserm U970, Paris Cardiovascular Research Center, Hôpital Européen Georges Pompidou Paris, France).

The data will be stored on a computer server dedicated only to the storage and processing of the project data. The computer used for the analyzes is in a locked room within the secure premises of the European Georges Pompidou Hospital ( INSERM U970, Cardiovascular Research Center of Paris), guarded 24/24 with access by name badge.

Persons having direct access (for example, investigators, persons in charge of quality control, Clinical Research Assistants, and all persons involved in the study) take all necessary precautions to ensure the confidentiality of information relating to the persons who are suitable for it. All the co-investigators will have access to the data of the study to develop their working hypotheses within the premises of the INSERM U970, but no data can be transferred outside the dedicated and secure computer server.

European George Pompidou Hospital as sponsor is subject to the rights and obligations as 'data controller' set forth under the General Data Protection Regulation 2016/679 ("GDPR") in relation to the processing of personal data in accordance with the protocol. Participating site is subject to the rights and obligations as 'data processor' set forth under the GDPR in relation to the processing of personal data in accordance with the protocol. Sponsor and participating site agree that such data: (a) is to be used only for the purposes as described in the protocol; (b) will not be used for commercial purposes and (c) will not be transferred to a third party. Sponsor and participating site shall provide sufficient safeguards in respect of the administrative, technical and organizational measures for processing personal data and take all necessary measures to protect the confidentiality, privacy and prevention from accidental or unauthorized destruction, accidental loss, as well as from alteration, access and any other unauthorized processing of the data. Participating site shall promptly inform Sponsor of any security breach, reasonably assist Sponsor with the handling of (a) responses to any security breach and (b) any requests from data subjects under Chapter III of the GDPR. The Participating site shall obtain prior specific or general written consent from Sponsor before engaging a subprocessor of the Personal Data. Participating site remains data controller of the data contained in its patients' medical records for the purposes of providing medical care to its patients and for other academic research purposes initiated by participating site.

3. Quality assurance:

1. Verification of data:

   Source data will be verified by comparing the data to medical records and case report forms in the form of a random sample.
2. Clinical events committee:

To avoid or minimize bias, an independent clinical events committee at the main investigational site, consisting of independent physicians, assesses all primary endpoint clinical events.

ELIGIBILITY:
Inclusion Criteria:

* patients >16 years of age
* sRV and a transposition of the great arteries (TGA or ccTGA) with "two-ventricle circulation"

Exclusion Criteria: congenital heart diaese with univentricular heart physiology

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All adult patients (>16 years of age) with sRV and "two-ventricles" circulation, i.e, patients with a transposition of the great arteries palliated by atrial switch procedure and patients with a congenitally corrected transposition of the great arteries, under active follow-up between January 1, 2000 and September 30, 2018
Sampling Method: Probability Sample
Enrollment: 1240 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
sudden cardiac death, | 2000 to 2018
near-miss sudden death | 2000 to 2018
sustained VT requiring defibrillation | 2000 to 2018

SECONDARY OUTCOMES:
all causes of death | 2000 to 2018
  heart failure, atrial arrhythmia, AV block, stroke

CONTACTS AND LOCATIONS:
Overall Officials: Magalie Ladouceur, Dr, Principal Investigator — Hopital Europeen Georges Pompidou
Locations (1):
- Hopital Europen Georges Pompidou, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kammeraad JA, van Deurzen CH, Sreeram N, Bink-Boelkens MT, Ottenkamp J, Helbing WA, Lam J, Sobotka-Plojhar MA, Daniels O, Balaji S. Predictors of sudden cardiac death after Mustard or Senning repair for transposition of the great arteries. J Am Coll Cardiol. 2004 Sep 1;44(5):1095-102. doi: 10.1016/j.jacc.2004.05.073. PMID 15337224
- [Result] Schwerzmann M, Salehian O, Harris L, Siu SC, Williams WG, Webb GD, Colman JM, Redington A, Silversides CK. Ventricular arrhythmias and sudden death in adults after a Mustard operation for transposition of the great arteries. Eur Heart J. 2009 Aug;30(15):1873-9. doi: 10.1093/eurheartj/ehp179. Epub 2009 May 22. PMID 19465439
- [Result] Khairy P, Harris L, Landzberg MJ, Fernandes SM, Barlow A, Mercier LA, Viswanathan S, Chetaille P, Gordon E, Dore A, Cecchin F. Sudden death and defibrillators in transposition of the great arteries with intra-atrial baffles: a multicenter study. Circ Arrhythm Electrophysiol. 2008 Oct;1(4):250-7. doi: 10.1161/CIRCEP.108.776120. Epub 2008 Sep 12. PMID 19808416